CLINICAL TRIAL: NCT01099072
Title: Carnitine as an Adjunct to Methylphenidate for the Treatment of Attention Deficit Hyperactivity Disorder Children and Adolescents in the Placebo Control Double -Blind Randomized Clinical Trail
Brief Title: Carnitine as an Adjunct to Methylphenidate for the Treatment of Attention Deficit Hyperactivity Disorder
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8642
Record Dates: First submitted 2010-04-03; First posted 2010-04-06 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; carnitine; methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylphenidate+placebo (Active Comparator): methylphenidate at a dose of 20-30 mg/day depending on weight (20 mg/day for <30 Kg and 30 mg/day for >30 Kg)+ Placebo
  Interventions: Drug: Methylphenidate+placebo
- methylphenidate+carnitine (Experimental)
  Interventions: Drug: methylphenidate+carnitine

INTERVENTIONS:
Drug: Methylphenidate+placebo — methylphenidate at a dose of 20-30 mg/day depending on weight (20 mg/day for <30 Kg and 30 mg/day for >30 Kg)+ Placebo
  Arms: Methylphenidate+placebo
Drug: methylphenidate+carnitine — methylphenidate at a dose of 20-30 mg/day depending on weight (20 mg/day for <30 Kg and 30 mg/day for >30 Kg)+ Carnitine 500-1500 mg/day (depending on weight )
  Arms: methylphenidate+carnitine

SUMMARY:
Attention-deficit hyperactivity disorder (ADHD) is the most common neurobehavioural disorder of childhood. The investigators hypothesized that carnitine would be beneficial for treatment of ADHD, and this could be evaluated in a double blind, randomized, parallel group comparison of carnitine+methylphenidate and methylphenidate +placebo.

This will be a six-week, parallel group, randomized clinical trial undertaken in an outpatient child and adolescent clinic at Roozbeh Psychiatric Hospital in Tehran, Iran during April 2010-May 2010.

40 male and female subjects, ages 6 to 17 years with a Diagnostic and Statistical Manual, Fourth Edition, Text Revision (DSM-IV-TR) diagnosis of ADHD will be study population of this trial. At screening, investigators conduct a psychiatric evaluation with the DSM-IV-TR criteria for ADHD and the Kiddie Schedule for Affective Disorders and Schizophrenia-Present and Lifetime diagnostic interview and perform a complete medical history and physical examination.

The diagnosis of ADHD will be confirmed by a child and adolescent psychiatrist before participants will be initiated into the study. All patients will be newly diagnosed. Parents were carefully interview and ask to rate the severity of the DSM-IV-TR ADHD symptoms that their children display at home. Children will be excluded if they have a history or current diagnosis of pervasive developmental disorders, schizophrenia or other psychiatric disorders(DSM-IV axis I); any current psychiatric comorbidity that required pharmacotherapy; any evidence of suicide risk and mental retardation (I.Q. <70). In addition, patients will be excluded if they have a clinically significant chronic medical condition, including organic brain disorder, seizures and, current abuse or dependence on drugs within 6 months. Additional exclusion criteria will be hypertension, hypotension. To participate, parents and children have to be willing to comply with all requirements of the study. After a description of the procedures and purpose of the study, written informed consent will be obtained from each patient's parent or guardian. Informed consent will receive before the administration of any study procedure or dispensing of study medication in accordance with the ethical standards of the investigative site's institutional review board and with the Helsinki declaration of 1975, as revised in 2000. The protocol will be approved by the Institutional Review Board (IRB) of Tehran University of Medical Sciences.

Patients will be randomized to receive a carnitine+methylphenidate and methylphenidate +placebo in a 1: 1 ratio using a computer-generated code.

All study subjects will be randomly assigned to receive treatment using methylphenidate at a dose of 20-30 mg/day depending on weight (20 mg/day for <30 Kg and 30 mg/day for >30 Kg)+ Carnitine 500-1500 mg/day (depending on weight ) or methylphenidate at a dose of 20-30 mg/day depending on weight (20 mg/day for <30 Kg and 30 mg/day for >30 Kg)+ Placebo for a 6 week double blind, randomized clinical.

The principal measure of outcome will be the Parent and Teacher ADHD Rating Scale-IV that has been used extensively in Iran in school-age children and provides valid measures of behavioral abnormality and attention trial.

Side effects will be systematically recorded throughout the study and will be assessed using a checklist that comprises 20 side effects including psychic, neurologic, autonomic and other side effects, administered by a child psychiatrist on days 7, 21and 42. Side effects, administered by a child psychiatrist on days 7, 21and 42.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of ADHD will be confirmed by a child and adolescent psychiatrist before participants will be initiated into the study.
* All patients will be newly diagnosed. Parents were carefully interview and ask to rate the severity of the DSM-IV-TR ADHD symptoms that their children display at home.

Exclusion Criteria:

* Children will be excluded if they have a history or current diagnosis of pervasive developmental disorders, schizophrenia or other psychiatric disorders(DSM-IV axis I)
* Any current psychiatric comorbidity that required pharmacotherapy
* Any evidence of suicide risk and mental retardation (intelligence quotient [I.Q.] <70).
* In addition, patients will be excluded if they have a clinically significant chronic medical condition, including organic brain disorder, seizures and, current abuse or dependence on drugs within 6 months.
* Additional exclusion criteria will be hypertension, hypotension.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The principal measure of outcome will be the Parent and Teacher ADHD Rating Scale-IV | 6 weeks
  Parent and Teacher ADHD Rating Scale-IV that has been used extensively in Iran in school-age children and provides valid measures of behavioral abnormality and attention trial.

CONTACTS AND LOCATIONS:
Overall Officials: Shahin Akhondzadeh, Ph.D., Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Tehran University of Medical Sciences, Tehran, Tehran Province, Iran